CLINICAL TRIAL: NCT04959123
Title: Does the Common Practice of Adding Diluted Epinephrine in Tranverse Abdominal Plan Block to Ropivacaine Significantly Decrease the Peak Systemic Resorption of Ropivacaine?
Acronym: ROPIVADRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-PP-28
Record Dates: First submitted 2021-06-28; First posted 2021-07-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-03

CONDITIONS: Bowel Disease
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine (Active Comparator): Patients receive 0.5 mg/kg of actual weight of ropivacaine; the appropriate dose of ropivacaine is drawn from an ampoule of 0.5% ropivacaine, i.e., 5 mg/mL (example for a 75 kg individual: 7.5 mL in each syringe) In the "Ropivacaine only" group, there is no adrenaline, the syringe loaded with ropivacaine is supplemented to 20 mL with a 0.9% sodium chloride solution
  Interventions: Other: pharmacokinetic analysis
- Ropivacaine + Epinephrine (Experimental): Patients receive 0.5 mg/kg of actual weight of ropivacaine; the appropriate dose of ropivacaine is drawn from an ampoule of 0.5% ropivacaine, i.e., 5 mg/mL (example for a 75 kg individual: 7.5 mLn each syringe) In the "ropivacaine + epinephrine" group, 0.1 mL of a 1 mg/mL ampoule of epinephrine is added to each syringe before making up to 20 mL (i.e., 100 µg of epinephrine for 20 mL of final solution, i.e., 5 µg/mL, i.e., 1 : 200000).
  Interventions: Other: pharmacokinetic analysis

INTERVENTIONS:
Other: pharmacokinetic analysis — Non-compartmental descriptive pharmacokinetic analysis (i.e. without the need for mathematical modelling), with determination of the pharmacokinetic parameters of interest either directly from the experimental points (Cmax, Tmax), or from simple mathematical equations (calculation of the area under the curve (AUC) by the trapezoidal method, calculation of the terminal slope of elimination)

SUMMARY:
Locoregional anesthesia techniques are now widely recommended in perioperative multimodal analgesia protocols. The transverse abdominal plane block (TAP block), which consists of the injection of a local anesthetic in the vascular-nervous plane between the internal oblique muscle and the transverse abdominal muscle, has seen a significant increase in abdominal surgery with the advent of ultrasound guidance. Aimed at blocking the nerves destined to the antero-lateral abdominal wall, it has shown a benefit in several abdominopelvic surgeries with in particular a reduction of pain and a morphine sparing during the 24 postoperative hours as well as a shortening of the delay of resumption of the intestinal transit.

Ropivacaine is the molecule of choice in transverse abdominal plane block because of its better safety profile among long-acting local anesthetics. Nevertheless, transverse abdominal plane block using ropivacaine has a risk of systemic toxicity, correlated to the peak systemic resorption of the local anesthetic, whose low incidence is probably underestimated in patients under general anesthesia.

In this context, the addition of diluted adrenaline to the ropivacaine solution is a common practice in loco-regional anesthesia, including transverse abdominal plane block, to increase the duration of the peripheral block and reduce the peak plasma concentration of the local anesthetic.

The objective of our study is to compare the pharmacokinetics of total and free ropivacaine administered in transverse abdominal plane block at the minimum effective dosage of 1 mg/kg without and with the addition of epinephrine at the concentration of 1:200000 (5 µg/mL) in patients scheduled for laparoscopic colectomy. The hypothesis is a significant reduction in the mean maximum concentration (Cmax) of total or free plasma ropivacaine in the adrenalized block transverse abdominal plane group.

The practical applications in case of verification of the hypothesis are the provision of an argument to recommend the systematic adrenalization of the transverse abdominal plane block with ropivacaine in the interest of patient safety and the prospect of a downward reassessment of the minimum time to be respected between the administration of a transverse abdominal plane block with ropivacaine and that of another locoregional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years) scheduled for laparoscopic colectomy
* Physical status score ( American Society of Anesthesiologists) ≤ 3
* Non-obese (Body Mass Index < 30)
* Affiliated with a social security plan
* Having signed an informed consent
* Normal preoperative electrocardiogram including, but not limited to, a non-extended QTc interval (< 0.45 s in men and < 0.47 s in women).

Exclusion Criteria:

* Presence of a contraindication for local anesthesia (injection site infection, coagulopathy)
* Known allergy to local anesthetics
* Known renal or hepatic insufficiency
* Pregnant or breastfeeding women
* Medical or psychiatric condition that makes communication difficult
* Chronic use of drugs that interfere with CYP1A2 metabolism of ropivacaine such as fluvoxamine (a potent CYP1A2 inhibitor)
* Chronic use of opioids or other treatments for chronic pain
* Chronic use of anti-arrhythmic drug(s) or drugs that can prolong the QTc space such as haloperidol, amiodarone, sotalol, etc.
* Protected persons defined in the following articles of the public health code:

L. 1121-6: persons deprived of liberty by a judicial or administrative decision, persons hospitalized without consent and persons admitted to a health or social institution for purposes other than research; L. 1121-8: adults subject to a legal protection measure or unable to express their consent; L. 1122-1-2: persons in emergency situations who are unable to give prior consent.

- Patients participating in other research involving the human person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-11-19 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Difference in mean peak concentrations (Cmax) of total and free plasma ropivacaine after transversus abdominis plane block between both groups | 240 minutes after transversus abdominis plane block
  Difference between the mean peak concentrations (Cmax) of total and free plasma ropivacaine after transversus abdominis plane block 1 mg/kg of both transversus abdominis plane block-adrenaline+ and transversus abdominis plane block-adrenaline- groups (before and 15, 30, 45, 60, 90, 120, 180, and 240 minutes after transversus abdominis plane block).

SECONDARY OUTCOMES:
Difference in mean Tmax of total and free plasma ropivacaine between the two groups | 240 minutes after transversus abdominis plane block
  Difference in mean Tmax (time to maximum concentration Cmax) of total and free plasma ropivacaine between the two groups transversus abdominis plane block-adrenaline+ and transversus abdominis plane block-adrenaline-
Efficacy markers : pain visual analog scale | 24 hours
  Collection of efficacy markers :pain visual analog scale. Score from 0 to 10. 0 being no pain and 10 being the maximum pain imaginable.
Efficacy markers : morphine consumption | 24 hours
  whether or not to use morphine during the 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Romain ROZIER, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de nice - Anesthésie Réanimation, Nice, Alpes-Maritimes, France

REFERENCES:
- [Derived] Rozier R, Le Guennec Y, Capdevila X, Le Louarn E, Balbo J, Lavrut T, Baque P, Perus O, Destere A, Maurice-Szamburski A. Impact of epinephrine on ropivacaine pharmacokinetics in TAP blocks: a randomized controlled trial. Reg Anesth Pain Med. 2025 Mar 17:rapm-2025-106500. doi: 10.1136/rapm-2025-106500. Online ahead of print. PMID 40096993